CLINICAL TRIAL: NCT02761174
Title: Topical Brimonidine Reduces IPL-induced Erythema Without Affecting Efficacy: a Randomized Controlled Trial in Patients With Facial Telangiectasias
Brief Title: Topical Brimonidine to Reduce Inflammation After IPL-treatment in Patients With Facial Telangiectasias
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Collaborators: Skinperium, Christine Dierickx (Unknown); Ellipse A/S Agern Allé 11, 2970 Hørsholm (Unknown)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Professor, MD, DMSc, PhD, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-004789-27
Record Dates: First submitted 2016-03-17; First posted 2016-05-04 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Telangiectasias
Keywords: Vascular lesions; inflammation; IPL
MeSH Terms: conditions — Telangiectasis; Inflammation | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brimonidine (Mirvaso cream) (Active Comparator): This is a split-face study, and patients are thereby their own control. Patients receive IPL-treatment and air-cooling to the whole face (control) and 0.5 g of brimonidine (Mirvaso cream) to the randomized side of the face.
  Interventions: Drug: Brimonidine
- IPL+air-cooling (Other): This is a split-face study, and patients are thereby their own control. Patients receive IPL-treatment and air-cooling to the whole face and IPL+air-cooling (control) are thereby compared to IPL+air-cooling+brimonidine (Mirvaso cream).
  Interventions: Other: IPL+air-cooling

INTERVENTIONS:
Drug: Brimonidine — Patients receive brimonidine to half of their face, whereas the other half receives no treatment and thereby patients are their own control
  Other Names: Mirvaso cream
  Arms: Brimonidine (Mirvaso cream)
Other: IPL+air-cooling — IPL+air-cooling are applied to the whole face and the control side thereby only receives IPL+air-cooling
  Arms: IPL+air-cooling

SUMMARY:
The aim of the study is to investigate whether brimonidine cream can reduce IPL-induced inflammation in terms of redness, swelling and pain in patients with facial vascular lesions (telangiectasias). Furthermore, the effect of brimonidine cream on IPL-efficacy is evaluated one month after final IPL-treatment.

The hypothesis is that brimonidine, which has been proved effective in reduction of symptomatic erythema in patients with rosacea, also may have the ability to reduce IPL-induced erythema. Since the potential reduction in erythema is caused by vasoconstriction, brimonidine may further reduce IPL-induced oedema and pain.

DETAILED DESCRIPTION:
Study design The study is designed as a dual-centre, randomized, intra-individual, split-face clinical controlled trial with blinded outcome assessment. A total of 20 patients with moderate to severe facial telangiectasias, without other clinical active dermatological disease in the skin, will be included. Severity and distribution (cheek, nose and chin) of telangiectasias must be symmetrical between facial sides in the individual patient at inclusion. All patients will receive IPL-treatments to both sides of the face. Before the first IPL-treatment, the left and right side of the face will be randomized to either brimonidine (Mirvaso) or only IPL-treatment and air-cooling (control), respectively. The study is conducted in an international collaboration between Bispebjerg Hospital, Department of Dermatology in Denmark and "Skinperium" private practice in Belgium.

Interventions Patients are asked to attend 3 treatment days and 2 follow-up visits. Treatment days are planed with 3 weeks intervals (± 5 days) and follow-up visits are planned at trial day 2 (one day after treatment day 1) and at 1 month (± 5 days) after the final treatment day. The consultations are estimated to last between half an hour and two hours. Patients are further asked to fill out patient diaries in the first 6 days after follow-up visit at trial day 2.

At each treatment day, patients receive 1) IPL of their whole face, 2) brimonidine is thereafter applied to the facial side randomized to treatment followed by 3) air-cooling, which is applied to the whole face of the patient in accordance with clinical guidelines.

Efficacy endpoints & evaluation methods

Primary efficacy endpoint:

To investigate whether topical brimonidine can reduce IPL-induced inflammatory response

Secondary efficacy endpoints:

1. IPL-induced treatment efficacy on telangiectasias with and without application of brimonidine
2. Patient-evaluated subjective discomfort and pain in the treatment area
3. Overall patient satisfaction

Primary efficacy endpoint is quantified by reduction in erythema and oedema assessed by blinded clinical on-site evaluation and by blinded photo-evaluation.

Secondary efficacy endpoints regarding point 1 are quantified by blinded photo-evaluation obtained with a Visia camera, in which baseline-photos are compared to photos from the final follow-up visit. Point 2 and 3 are evaluated on two separate 0-10 point Visual Analogue Scales (VAS) on discomfort/pain and patient satisfaction, respectively. Patient satisfaction is further evaluated in patient diaries.

Product Mirvaso® (brimonidine tartrate (3,3mg/1g), Galderma Nordic) One gram of gel contains 3.3 mg of brimonidine, equivalent to 5 mg of brimonidine tartrate.

Excipient(s) with known effect:

One gram of gel contains 1 mg methylparahydroxybenzoate (E218) and 55 mg propylene glycol.

Other excipients:

* Carbomer Methylparahydroxybenzoate (E218) Phenoxyethanol
* Glycerol
* Titanium dioxide
* Propylene glycol
* Sodium hydroxide
* Purified water

Statistic analysis Primary efficacy endpoint is difference in inflammation between brimonidine vs. control.

Wilcoxon signed-rank test will be used for paired comparison to evaluate eventual differences between brimonidine vs. control. Analysis on Per-Protocol will only include the patients completing the study according to protocol.

Sample size Estimation of sample size is based on clinical on-site evaluation on inflammation 30 minutes after incubation of brimonidine (effect of brimonidine is evident after 30 minutes cf.´Summary of Product Characteristics) and 24 hours after application.

With a power of 90%, a type I error probability of 5% and an estimated standard deviation of 25%, we should include 17 patients to detect a minimum relevant difference (MIREDIF) of 20% between brimonidine and control. We choose a 20% MIREDIF, since a reduction in inflammation <20%, based on a resource economic point of view is considered clinical irrelevant. Based on earlier experience and duration of the trial, a 15% dropout rate should be taken into account and therefore, a total of 20 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe facial telangiectasias referred to laser or IPL-treatment. Severity and distribution of telangiectasias must be symmetrical between left and right side of the face in the individual patient
* Telangiectasias may be observed in connection with rosacea, but rosacea must not demonstrate clinical active inflammation or acne
* 18-65 years of age
* Fitzpatrick skin type I-III
* Fertile women must document non-reactive urine pregnancy test at the day of inclusion
* During the study, fertile women must be using effective birth control. Effective contraception is defined as follows:

  * Injectable, implantable or orally taken hormones;
  * Intrauterine device;
  * Trans-abdominal surgical sterilization;
  * Sterilization implant device;
  * Surgical sterilization of male partner;
  * Complete abstinence from sexual intercourse for two weeks before exposure to study medication and throughout the clinical study
* Verbal and written consent to participate in the study
* Documentation of medicine status

Exclusion Criteria:

* Clinical active dermatological disease in the face
* Wounds, dermatitis, tattoos or scars in treatment area
* Allergies to ingredients in Mirvaso
* Current treatment with monoamine oxidase inhibitors, tricyclic or tetracyclic antidepressants which interacts with the noradrenergic transmission
* Current treatment with other systemic adrenergic receptor agonists or antagonists
* Patients with known liver or renal disease
* UV-exposure (solarium or sunbathing) or other treatment within the last month that enhances skin pigmentation
* Use of other topical agents that may interact with treatment
* Local or systemic treatment with photosensitizing drugs
* Pregnancy and breastfeeding women
* Current participation in other clinical trials
* Patients that are considered incapable of complying with the protocol, i.e. patients suffering from dementia, alcoholism or psychiatric conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-13 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Reduction in erythema quantified by blinded clinical on-site evaluation and by blinded photo-evaluation. | Throughout the study, a period of 10 weeks
  Erythema is evaluated on the international validated, "Clinician's Erythema Assessment" (CEA) 5-point scale:
  0, Clear Clear skin with no signs of erythema
  1. Almost clear Almost clear; slight redness
  2. Mild Mild erythema; definite redness
  3. Moderate Moderate erythema; marked redness
  4. Severe Severe erythema; fiery redness
Reduction in oedema quantified by blinded clinical on-site evaluation and by blinded photo-evaluation. | Throughout the study, a period of 10 weeks
  Oedema is evaluated on a 4-point scale: 0 = no oedema, 1 = little oedema, 2 = moderate oedema and 3 = severe oedema.

SECONDARY OUTCOMES:
The effect of brimonidine on IPL-efficacy quantified by blinded photo-evaluation obtained with a Visia camera, in which baseline-photos are compared to photos from the final follow-up visit. | At the end of the study (after 10 weeks)
  Baseline photos are compared to photos at final follow-up visit approximate 10 weeks after.
Patient discomfort and pain | Throughout the study, a period of 10 weeks
  Patient discomfort and pain are evaluated on a numeric Visual Analogue Scale (VAS) from 0 (no discomfort/pain) to 10 (extreme discomfort/pain) separately for brimonidine and control
Patient overall satisfaction | Throughout the study, a period of 10 weeks
  Patients evaluate their overall satisfaction with brimonidine to reduce IPL-induced inflammation on a numeric VAS from 0 (poor outcome) to 10 (excellent outcome). Inflammation is described as redness, swelling and pain to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, Prof., MD, Principal Investigator — Department of Dermatology
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Sponsor and investigator allow access to registries, CRF and trial master files in case of audit or quality inspection from relevant authorities such as GCP-unit, Danish Health and Medicine Authority or The Regional Committee on Health Research Ethics

REFERENCES:
- [Background] Tierney E, Hanke CW. Randomized controlled trial: Comparative efficacy for the treatment of facial telangiectasias with 532 nm versus 940 nm diode laser. Lasers Surg Med. 2009 Oct;41(8):555-62. doi: 10.1002/lsm.20811. PMID 19746429
- [Background] Adamic M, Pavlovic MD, Troilius Rubin A, Palmetun-Ekback M, Boixeda P. Guidelines of care for vascular lasers and intense pulse light sources from the European Society for Laser Dermatology. J Eur Acad Dermatol Venereol. 2015 Sep;29(9):1661-78. doi: 10.1111/jdv.13177. Epub 2015 Apr 30. PMID 25931003
- [Background] Taub AF, Devita EC. Successful treatment of erythematotelangiectatic rosacea with pulsed light and radiofrequency. J Clin Aesthet Dermatol. 2008 May;1(1):37-40. PMID 21103309
- [Background] Tanghetti EA. Split-face randomized treatment of facial telangiectasia comparing pulsed dye laser and an intense pulsed light handpiece. Lasers Surg Med. 2012 Feb;44(2):97-102. doi: 10.1002/lsm.21151. Epub 2011 Dec 16. PMID 22180317
- [Background] Nymann P, Hedelund L, Haedersdal M. Long-pulsed dye laser vs. intense pulsed light for the treatment of facial telangiectasias: a randomized controlled trial. J Eur Acad Dermatol Venereol. 2010 Feb;24(2):143-6. doi: 10.1111/j.1468-3083.2009.03357.x. PMID 20205349
- [Background] Uebelhoer NS, Bogle MA, Stewart B, Arndt KA, Dover JS. A split-face comparison study of pulsed 532-nm KTP laser and 595-nm pulsed dye laser in the treatment of facial telangiectasias and diffuse telangiectatic facial erythema. Dermatol Surg. 2007 Apr;33(4):441-8. doi: 10.1111/j.1524-4725.2007.33091.x. PMID 17430378
- [Background] Papageorgiou P, Clayton W, Norwood S, Chopra S, Rustin M. Treatment of rosacea with intense pulsed light: significant improvement and long-lasting results. Br J Dermatol. 2008 Sep;159(3):628-32. doi: 10.1111/j.1365-2133.2008.08702.x. Epub 2008 Jun 28. PMID 18565174
- [Background] Clark C, Cameron H, Moseley H, Ferguson J, Ibbotson SH. Treatment of superficial cutaneous vascular lesions: experience with the KTP 532 nm laser. Lasers Med Sci. 2004;19(1):1-5. doi: 10.1007/s10103-004-0294-x. Epub 2004 Apr 14. PMID 15316851
- [Background] Eremia S, Li CY. Treatment of face veins with a cryogen spray variable pulse width 1064 nm Nd:YAG Laser: a prospective study of 17 patients. Dermatol Surg. 2002 Mar;28(3):244-7. doi: 10.1046/j.1524-4725.2002.01217.x. PMID 11896777
- [Background] Bjerring P, Christiansen K, Troilius A. Intense pulsed light source for treatment of facial telangiectasias. J Cosmet Laser Ther. 2001 Dec;3(4):169-73. doi: 10.1080/14764170160260744. PMID 12554324
- [Background] Mark KA, Sparacio RM, Voigt A, Marenus K, Sarnoff DS. Objective and quantitative improvement of rosacea-associated erythema after intense pulsed light treatment. Dermatol Surg. 2003 Jun;29(6):600-4. doi: 10.1046/j.1524-4725.2003.29141.x. PMID 12786702
- [Background] Anderson RR, Parrish JA. Selective photothermolysis: precise microsurgery by selective absorption of pulsed radiation. Science. 1983 Apr 29;220(4596):524-7. doi: 10.1126/science.6836297.
- [Background] Srinivas CR, Kumaresan M. Lasers for vascular lesions: standard guidelines of care. Indian J Dermatol Venereol Leprol. 2011 May-Jun;77(3):349-68. doi: 10.4103/0378-6323.79728. PMID 21508585
- [Background] Handley JM. Adverse events associated with nonablative cutaneous visible and infrared laser treatment. J Am Acad Dermatol. 2006 Sep;55(3):482-9. doi: 10.1016/j.jaad.2006.03.029. PMID 16908355
- [Background] Alam M, Omura NE, Dover JS, Arndt KA. Clinically significant facial edema after extensive treatment with purpura-free pulsed-dye laser. Dermatol Surg. 2003 Sep;29(9):920-4. doi: 10.1046/j.1524-4725.2003.29254.x. PMID 12930333
- [Background] Lou WW, Quintana AT, Geronemus RG, Grossman MC. Effects of topical vitamin K and retinol on laser-induced purpura on nonlesional skin. Dermatol Surg. 1999 Dec;25(12):942-4. doi: 10.1046/j.1524-4725.1999.99145.x. PMID 10594627
- [Background] Leu S, Havey J, White LE, Martin N, Yoo SS, Rademaker AW, Alam M. Accelerated resolution of laser-induced bruising with topical 20% arnica: a rater-blinded randomized controlled trial. Br J Dermatol. 2010 Sep;163(3):557-63. doi: 10.1111/j.1365-2133.2010.09813.x. PMID 20412090
- [Background] Alonso D, Lazarus MC, Baumann L. Effects of topical arnica gel on post-laser treatment bruises. Dermatol Surg. 2002 Aug;28(8):686-8. doi: 10.1046/j.1524-4725.2002.02011.x. PMID 12174058
- [Background] Oge' LK, Muncie HL, Phillips-Savoy AR. Rosacea: Diagnosis and Treatment. Am Fam Physician. 2015 Aug 1;92(3):187-96. PMID 26280139
- [Background] Benkali K, Leoni M, Rony F, Bouer R, Fernando A, Graeber M, Wagner N. Comparative pharmacokinetics and bioavailability of brimonidine following ocular and dermal administration of brimonidine tartrate ophthalmic solution and gel in patients with moderate-to-severe facial erythema associated with rosacea. Br J Dermatol. 2014 Jul;171(1):162-9. doi: 10.1111/bjd.12881. Epub 2014 Jul 16. PMID 24506775
- [Background] Piwnica D, Rosignoli C, de Menonville ST, Alvarez T, Schuppli Nollet M, Roye O, Jomard A, Aubert J. Vasoconstriction and anti-inflammatory properties of the selective alpha-adrenergic receptor agonist brimonidine. J Dermatol Sci. 2014 Jul;75(1):49-54. doi: 10.1016/j.jdermsci.2014.04.002. Epub 2014 Apr 16. PMID 24802713
- [Background] Fowler J, Jarratt M, Moore A, Meadows K, Pollack A, Steinhoff M, Liu Y, Leoni M; Brimonidine Phase II Study Group. Once-daily topical brimonidine tartrate gel 0.5% is a novel treatment for moderate to severe facial erythema of rosacea: results of two multicentre, randomized and vehicle-controlled studies. Br J Dermatol. 2012 Mar;166(3):633-41. doi: 10.1111/j.1365-2133.2011.10716.x. PMID 22050040
- [Background] Fowler J, Tan J, Jackson JM, Meadows K, Jones T, Jarratt M, Leoni M; Brimonidine Phase III Study Group. Treatment of facial erythema in patients with rosacea with topical brimonidine tartrate: correlation of patient satisfaction with standard clinical endpoints of improvement of facial erythema. J Eur Acad Dermatol Venereol. 2015 Mar;29(3):474-81. doi: 10.1111/jdv.12587. Epub 2014 Jul 30. PMID 25074756
- [Background] van Zuuren EJ, Fedorowicz Z. Interventions for rosacea: abridged updated Cochrane systematic review including GRADE assessments. Br J Dermatol. 2015 Sep;173(3):651-62. doi: 10.1111/bjd.13956. Epub 2015 Aug 30. PMID 26099423
- [Background] Johnson AW, Johnson SM. The Role of Topical Brimonidine Tartrate Gel as a Novel Therapeutic Option for Persistent Facial Erythema Associated with Rosacea. Dermatol Ther (Heidelb). 2015 Sep;5(3):171-81. doi: 10.1007/s13555-015-0078-1. Epub 2015 Jun 26. PMID 26112098
- [Background] Holmes AD, Waite KA, Chen MC, Palaniswamy K, Wiser TH, Draelos ZD, Rafal ES, Werschler WP, Harvey AE. Dermatological Adverse Events Associated with Topical Brimonidine Gel 0.33% in Subjects with Erythema of Rosacea: A Retrospective Review of Clinical Studies. J Clin Aesthet Dermatol. 2015 Aug;8(8):29-35. PMID 26345379
- [Background] Moore A, Kempers S, Murakawa G, Weiss J, Tauscher A, Swinyer L, Liu H, Leoni M. Long-term safety and efficacy of once-daily topical brimonidine tartrate gel 0.5% for the treatment of moderate to severe facial erythema of rosacea: results of a 1-year open-label study. J Drugs Dermatol. 2014 Jan;13(1):56-61. PMID 24385120
- See also: European Medicines Agency — http://ec.europa.eu/health/documents/community-register/2014/20140221127901/anx_127901_en.pdf